CLINICAL TRIAL: NCT03876548
Title: Initial Assessment of a Topical Cadexomer Iodine Gel Efficacy on Keloid Scar Revision: A Pilot Clinical Study
Brief Title: Initial Assessment of a Topical Cadexomer Iodine Gel Efficacy on Keloid Scar Revision
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Recruitment Challenges
Sponsor: Next Science TM (Industry)
Collaborators: Jacksonville Center For Clinical Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CSP-008
Record Dates: First submitted 2019-03-12; First posted 2019-03-15 (Actual); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Keloid Scar Following Surgery
Keywords: keloid
MeSH Terms: conditions — Keloid

STUDY DESIGN:
Intervention Model Description: Pilot study
Masking Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Cadexomer Iodine Gel (Experimental): Patients willy apply product to treatment site every other day for the next 28 days and cover with dressing or bandage.
  Interventions: Device: Cadexomer Iodine Gel

INTERVENTIONS:
Device: Cadexomer Iodine Gel — Subjects will apply gel product to keloid scar site every other day for 28 days following keloid scar revision surgery.

SUMMARY:
This is a 6 month, single site, interventional, open label prospective clinical study to evaluate the effects of a cadexomer iodine gel on the prevention of recurrent keloid formation in patients undergoing keloid scar revision.

DETAILED DESCRIPTION:
The objective of this 6 month, interventional, open label prospective pilot study is to evaluate the effects of a cadexomer iodine gel on the prevention of recurrent keloid formation in patients undergoing keloid scar revision. Adults 18 years and older with an established diagnosis of keloid scar formation, scheduled to undergo keloid scar revision surgery, and who meet the protocol's inclusion and exclusion criteria are eligible for this study. There will be a minimum of 20 completed subjects with up to 30 enrolled. After keloid revision surgery, subjects will apply product every other day for one month. There will be a total of 5 study visits: Visit 0 (Revision Surgery Date and Start of Treatment); Visit 1 (1 Week Post-Revision); Visit 2 (4 Weeks Post-Revision); Visit 3 (12 Weeks Post Revision); and Visit 4 (24 Weeks Post-Revision and Study Exit). Imaging, Patient and Observer Scar Assessment Scale questionnaires, and Dermatological Life Quality Index Questions will be collected. It is hypothesized that there will be a measurable reduction in the amount (number, size) of keloid formation and/or recurrence at 4, 12, and 24 weeks post revision surgery time points. The change in subjects' quality of life as measured by the the Dermatology Quality of Life Index will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

Each subject must meet the following criteria to be enrolled in this trial:

1. Male or female 18 years or older
2. Subject is healthy, as determined by the investigator based on a medical evaluation and history
3. Subject has an established diagnosis of keloid scar formation
4. Subject's keloid is on the arm or chest but not on the wrist, elbow, or antecubital fossa
5. Subject has one or more keloids eligible for scar revision
6. Subject has a keloid of appropriate size (1 to 2.5 cm in length, 4 to 5 mm in width, and 3 to 4 mm in height)
7. Subject has no known allergies to study products
8. Subject is willing and able to avoid total body water exposure from large bodies of water such as pools, lakes, oceans, etc. while using study medication
9. Subject is willing and able to comply with the requirements of the protocol
10. Subject is male or non-pregnant, non-lactating woman. Women must be one of the following:

    * Naturally postmenopausal defined as ≥1 year without menses and:

      * ≥ 55 years or
      * < 55 years with follicle-stimulating hormone (FSH)≥40.0 IU/L, or
    * Surgically sterile including hysterectomy, bilateral oophorectomy, and/or tubal ligation, or
    * Women of childbearing potential willing to use an acceptable method(s) of birth control during the study, while using study medication including:

      * Oral, topical, injectable, or implantable birth control medications,
      * Placement of an intrauterine device with or without hormones,
      * Barrier methods including condoms or occlusive cap with spermicidal foam or spermicidal jelly
      * Vasectomized male partner who is the sole partner for this patient
      * True abstinence that is in line with the preferred and usual lifestyle of the patient (periodic abstinence [eg, calendar, ovulation, symptothermal, postovulation methods], declaration of abstinence for the duration of the study or withdrawal are not acceptable methods of true abstinence).
    * There are no protocol-specific birth control requirements for men with partners who are able to become pregnant
11. Subject has understood and signed an Informed Consent Form

Exclusion Criteria:

Each subject must meet the following criteria to be enrolled in this trial:

1. Subject has an underlying known disease, a surgical or medical condition that in the opinion of the investigator might put the subject at risk
2. Subject's keloid scar is on the wrist, elbow, or antecubital fossa.
3. Subject is pregnant or breastfeeding at the time of enrollment or is planning to become pregnant at any point during the study period
4. Subject has a past history of coagulopathy
5. Subject has an underlying dermatological disease that in the opinion of the investigator could interfere with the study evaluations
6. Subject is treated with anticoagulants or antiplatelet therapies
7. Subject has a known allergy or sensitivity to any local anesthetic (such as lidocaine) or a local topical antiseptic that may be used (such as iodine)
8. Subject has known allergic reaction to the study product
9. Subject has a known history of shellfish allergy or sensitivity
10. Subject has known history of Hashimoto's Thyroiditis, Graves' disease, a thyroid disorder, a non-toxic goiter
11. Subject is taking Lithium, Sulphafurazoles or Sulphonylureas
12. Subject is prone to Vasovagal syncope
13. Subject is unable to provide signed and dated informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-02-07 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Scar measurement with Silhouette Camera Imaging | 24 weeks
  The keloid or keloid scar will measured using the Silhouette Camera Imaging System
Patient and Observer Scar Assessment Scale (Subject facing) | 24 weeks
  Patient and Observer Scar Assessment to be completed by the subject with the physician.
Patient and Observer Scar Assessment Scale (Non-Subject facing) | 24 weeks
  Patient and Observer Scar Assessment to be completed by the physician only.
Response Rate calculation | 24 weeks
  Response Rate calculation = Complete Remission + Partial Response (RR= CR + PR)

SECONDARY OUTCOMES:
Dermatology Quality of Life Index | 24 Weeks
  Dermatology Quality of Life Index Questionaire

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bernhardt, MD, Principal Investigator — Jacksonville Center For Clinical Research
Locations (1):
- Jacksonville Center for Clinical Research, Jacksonville, Florida, United States